CLINICAL TRIAL: NCT02828384
Title: Comparing the Effectiveness of Two Dietary Interventions for Fecal Incontinence: a Randomized, Controlled Trial.
Brief Title: Comparing the Effectiveness of Two Dietary Interventions for Fecal Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: The Rome Foundation (Unknown)
Responsible Party: Principal Investigator, Stacy Menees, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00079064
Record Dates: First submitted 2016-04-25; First posted 2016-07-11 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Fecal Incontinence
Keywords: fodmap diet
MeSH Terms: conditions — Fecal Incontinence | interventions — FODMAP Diet; Psyllium

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- low fodmap diet (Active Comparator): Subjects receive formalized teaching in low fodmap diet by a dietician
  Interventions: Other: low fodmap diet
- psyllium (Active Comparator): subjects receive 7.1 g of psyllium daily
  Interventions: Dietary Supplement: Psyllium

INTERVENTIONS:
Other: low fodmap diet — dietary teaching
  Arms: low fodmap diet
Dietary Supplement: Psyllium — 7.1g of psyllium daily
  Arms: psyllium

SUMMARY:
Background:

Fecal incontinence (FI) is a common complaint, and is often associated with diarrhea and urgency. Foods that are high in fermentable oligo-, di-, and mono-saccharides and polyols (FODMAPs) cause symptoms of diarrhea and urgency. Thus, assessing the impact of a low FODMAP diet in FI patients is needed.

Aims:

1. Compare the treatment response with a low FODMAP vs. psyllium based on number of episodes in patients with FI.
2. Compare the efficacy of a low FODMAP diet vs. psyllium in patients with FI on pre-specified clinical and quality of life endpoints.

Methods:

This is a prospective, randomized control trial of adults meeting the Rome III criteria for FI and at least 1 episode of FI due to loose stool per week. After a 2 week screening period and randomization, during which the severity of symptoms will be assessed and eligibility determined, patients will be randomized to psyllium vs. low FODMAP diet for 4 weeks. A total of 20 patients will be recruited for each arm.

The primary endpoint will be treatment response based on number of incontinence episodes. A treatment response is defined as a reduction in the number of FI episodes/week.

ELIGIBILITY:
Inclusion Criteria

1. Experience at least 1 episode/week of unintentional loss of stool associated with diarrhea/loose stool (Bristol stool scale of 5 or greater).
2. Subjects aged 18 and older meeting the Rome III criteria for Functional Fecal incontinence diagnostic criteria:

Recurrent uncontrolled passage of fecal material in an individual and one or more of the following:

1. Abnormal functioning of normally innervated and structurally intact muscles
2. Minor abnormalities of sphincter structure and/or innervation
3. Normal or disordered bowel habits, (i.e., diarrhea) Criteria fulfilled for the last 3 months

Exclusion Criteria

1. Abnormal innervation caused by lesion(s) within the brain (e.g., dementia), spinal cord, or sacral nerve roots, or mixed lesions (e.g., multiple sclerosis), or as part of a generalized peripheral or autonomic neuropathy
2. Anal sphincter abnormalities associated with a multisystem disease (e.g., scleroderma)
3. Structural or neurogenic abnormalities believed to be the major or primary cause of fecal incontinence
4. Have cognitive dysfunction or unable to understand or provide written informed consent
5. Pregnancy
6. FI with solid stool only
7. Comorbid medical problems that may affect gastrointestinal transit or motility: Inflammatory bowel disease, Extraintestinal disease known to affect the gastrointestinal system (i.e., scleroderma, unstable thyroid disease, etc.),Severe renal or hepatic disease
8. Previous abdominal surgery other than appendectomy, cholecystectomy, and gynecologic/urologic surgery.
9. . Previous treatment with low FODMAP diet.
10. Concurrent medications not permitted including probiotics, antibiotics, and narcotics.
11. Active participation in another form of dietary therapy.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-10-02 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in number of FI episodes from baseline to week 4 | 4 weeks from baseline
  Will compare baseline number of FI episodes to number of FI episodes at week 4

SECONDARY OUTCOMES:
number of people responding with decreased score in stool consistency | 4 week span from baseline
  For stool consistency, a responder with improvement will be defined as one who reports a decrease in mean daily BSFS value ( on a scale of 1-7 with 7 being watery stool) of 1 or more compared to baseline for ≥2 of 4 treatment weeks. The proportion of responders between the 2 groups will be compared.
number of people responding with reduction in stool frequency | 4 weeks from baseline
  The number of bowel movements will be recorded each day. Mean daily stool frequency will be averaged for each treatment group at baseline and weekly through week 4. These averages will be compared for the two groups.
Change in stool wet weight | 4 weeks from baseline
  The difference in stool mean wet weight between baseline and during week 4 will be calculated. The change from baseline for each group will be compared.
Change in Fecal incontinence severity index (FISI) | 4 weeks from baseline
  Compare baseline fecal incontinence severity index with 4 week FISI score.
Change in Fecal incontinence quality of life measure (FIqol) | 4 weeks from baseline
  Compare baseline fecal incontinence quality of life with 4 week Fiqol score
Change in Short Form Health survey-36 | 4 weeks from baseline
  Compare baseline generalized QOL with 4 week SF-36
Number of participants with reduction in fecal incontinence episodes of ≥50% during weeks 3 & 4 of each diet compared with baseline | 4 weeks from baseline
  Responders are those participants with a reduction in FI episodes of > 50%. The reduction will be measured by the change in mean number of episodes in week 3 and 4 (averaged) from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Stacy B Menees, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Menees SB, Jackson K, Baker JR, Fenner DE, Eswaran S, Nojkov B, Saad R, Lee AA, Chey WD. A Randomized Pilot Study to Compare the Effectiveness of a Low FODMAP Diet vs Psyllium in Patients With Fecal Incontinence and Loose Stools. Clin Transl Gastroenterol. 2022 Feb 19;13(3):e00454. doi: 10.14309/ctg.0000000000000454. PMID 35060943